CLINICAL TRIAL: NCT00422838
Title: Impact of Immune Responses in Chronic Hepatitis C Genotype 1,2,3 Virus Infected Patients During Treatment With Pegylated Interferon-alpha-2b and Ribavirin (CIRES).
Brief Title: Study Investigating Immunological Effects of Treatment for Chronic Hepatitis C Patients.
Acronym: CIRES
Status: Completed | Type: Observational
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Other Study IDs: CIRES
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis C; Liver; Immunology; Regulation
Keywords: Hepatitis C; Liver; immunology; regulation; Genotype 1,2,3; Treatment; Chronic; Pegylated interferon; Ribavirin
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC Serum RNA Liver infiltrating lymphocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Chronic HCV Genotype 1 monoinfection, never had interferon and ribavirin treatment
  Interventions: Procedure: fine-needle aspiration biopsy
- 2: Chronic HCV Genotype 2 or 3 monoinfection,never had interferon and ribavirin treatment
  Interventions: Procedure: fine-needle aspiration biopsy

INTERVENTIONS:
Procedure: fine-needle aspiration biopsy — aspiration of intrahepatic cells

SUMMARY:
Aim

To evaluate the effects of peginterferon and ribavirin therapy on the immune response in chronic HCV genotype 1,2 or 3 patients before, during and after treatment.

Background

Treatment of chronic hepatitis C (HCV) has shown a remarkable success. However, genotype 1 patients have reduced response rates. A better understanding and improvement of these results can now be considered the greatest challenge.

In chronically infected patients, HCV-specific immune responses are generally weak, narrowly focused, and often dysfunctional. The presence of HCV-specific cells suppressing the immune response (regulatory T-lymphocytes=Treg) are able to suppress the immune response. These Treg are possibly responsible for the impaired immune response.

Previous studies have indicated increased Treg frequency and activity of immune regulating mechanisms, locally in the liver, as a result of HCV re-infection. Hence, these Data highlight the importance of monitoring intrahepatic immune responses in addition to peripheral immune responses. Using the minimally-invasive technique of fine-needle aspiration biopsy (FNAB), it is now possible to obtain safe and frequent liver samples to monitor local antiviral immune responses in chronic HCV patients during antiviral therapy.

Rationale and hypothesis of the study

Our previous studies and current literature support the concept that Treg may contribute to HCV persistence by suppressing HCV-spec immune responses. The current study is designed to examine if peginterferon and ribavirin therapy affects the activity of Treg and DC, and if this results in enhanced HCV-specific immune responses.

Design

Single centre, translational and observational open label study with one arm of 20 genotype 1 patients and one arm of 7 genotype 2/3 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18-70 years of age, with evidence of a chronic hepatitis C - Genotype 1,2 or 3 infection.
* No previous treatment with, peginterferon or conventional interferon plus ribavirin combination therapy.
* Indication for antiviral therapy of hepatitis C according to current clinical guidelines.
* Written informed consent.

Exclusion Criteria:

* History or other evidence of severe illness, malignancy or any other condition which would make the patient, in the opinion of the investigators, unsuitable for the study.
* Presence of contra-indications for antiviral therapy with peginterferon or ribavirin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients chronically infected with HCV-genotype 1,2 or 3
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R.J. de Knegt, MD, PhD, Principal Investigator — Department of Gastroenterology & Hepatology - Erasmus Medical Center Rotterdam; H.L.A. Janssen, MD, PhD, Principal Investigator — Department of Gastroenterology & Hepatology - Erasmus Medical Center Rotterdam
Locations (1):
- Department of Gastroenterology & Hepatology, Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- See also: website of the Erasmus Medical Center Rotterdam — http://www.erasmusmc.nl
- See also: website of the Department of Gastroenterology & Hepatology - Erasmus Medical Center Rotterdam — http://www.gastrolab.nl/